CLINICAL TRIAL: NCT06849947
Title: Randomized Phase II Trial of Fulvestrant With Ribociclib Versus Physician's Choice Treatments for the Patients Who Recurred After Completion of Adjuvant Cyclin-Dependent Kinase 4/6 Inhibitors in HR+, HER2- Metastatic Breast Cancer as First Line Treatment (CLEE011AKR06R)
Brief Title: Fulvestrant With Ribociclib Versus Physician's Choice Treatments Recurred After Completion of Adjuvant Cyclin-Dependent Kinase 4/6 Inhibitors in HR+, HER2- Metastatic Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yeon Hee Park (Other)
Responsible Party: Sponsor-Investigator, Yeon Hee Park, Professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-02-104
Record Dates: First submitted 2025-02-23; First posted 2025-02-27 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer Metastatic
MeSH Terms: interventions — ribociclib; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ribociclib group (Experimental): ▪ Ribociclib group
  - Ribociclib (600 mg orally once daily on days 1 to 21 in a 28 day cycle) + Fulvestrant (500mg intramuscular injection on day 1 in a 28 day cycle and day 15 of Cycle 1) ± Leuprorelin (3.75 mg subcutaneously every 28 days in premenopausal or perimenopausal women)
  Interventions: Drug: Ribociclib with fulvestrant
- Physician's choice treatments group (Active Comparator): ▪ Fulvestrant or exemestane group
  1. Fulvestrant (500mg intramuscular injection on day 1 in a 28 day cycle and day15 of Cycle 1) ± Leuprorelin (3.75 mg subcutaneously every 28 days in premenopausal or periomenopausal women) OR,
  2. Exemestane (25 mg orally once daily on day 1 to 28 in a 28 day cycle) + Everolimus (10 mg orally once daily on day 1 to 28 in a 28 day cycle) ± Leuprorelin (3.75 mg subcutaneously every 28 days in premenopausal or perimenopausal women)
  Interventions: Drug: Physician's choice treatments group

INTERVENTIONS:
Drug: Ribociclib with fulvestrant — ▪ Ribociclib group
  - Ribociclib (600 mg orally once daily on days 1 to 21 in a 28 day cycle) + Fulvestrant (500mg intramuscular injection on day 1 in a 28 day cycle and day 15 of Cycle 1) ± Leuprorelin (3.75 mg subcutaneously every 28 days in premenopausal or perimenopausal women)
  Arms: Ribociclib group
Drug: Physician's choice treatments group — ▪Fulvestrant or exemestane group
  1. Fulvestrant (500mg intramuscular injection on day 1 in a 28 day cycle and day15 of Cycle 1) ± Leuprorelin (3.75 mg subcutaneously every 28 days in premenopausal or periomenopausal women) OR,
  2. Exemestane (25 mg orally once daily on day 1 to 28 in a 28 day cycle) + Everolimus (10 mg orally once daily on day 1 to 28 in a 28 day cycle) ± Leuprorelin (3.75 mg subcutaneously every 28 days in premenopausal or perimenopausal women)
  Arms: Physician's choice treatments group

SUMMARY:
▪ Fulvestrant With Ribociclib versus Physician's choice treatments for the patients who recurred after completion of Adjuvant Cyclin-Dependent Kinase 4/6 Inhibitors in HR+, HER2- Metastatic Breast Cancer as first line treatment

DETAILED DESCRIPTION:
1. Treatment Arm :

   Ribociclib (600 mg orally once daily on days 1 to 21 in a 28 day cycle) + Fulvestrant (500mg intramuscular injection on day 1 in a 28 day cycle and day 15 of Cycle 1) ± Leuprorelin (3.75 mg subcutaneously every 28 days in premenopausal or perimenopausal women) OR,
2. Control Arm (Physician's choice treatments)

   1. Fulvestrant (500mg intramuscular injection on day 1 in a 28 day cycle and day15 of Cycle 1) ± Leuprorelin (3.75 mg subcutaneously every 28 days in premenopausal or periomenopausal women) OR,
   2. Exemestane (25 mg orally once daily on day 1 to 28 in a 28 day cycle) + Everolimus (10 mg orally once daily on day 1 to 28 in a 28 day cycle) ± Leuprorelin (3.75 mg subcutaneously every 28 days in premenopausal or perimenopausal women)

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be at least 19 years of age at the time of signing the informed consent.
2. Patient has advanced (locoregionally recurrent or metastatic) breast cancer not amenable to curative therapy.
3. Patient has HR-positive/HER2-negative invasive breast cancer (based on most recently analyzed biopsy)

   1. HER2 status is defined as a negative in situ hybridization test or an IHC status of 0, 1+ or 2+. If IHC is 2+, a negative in situ hybridization (FISH, CISH, or SISH) test is required by local laboratory testing, according to ASCO/CAP guidelines for HER2 testing (Wolff et al. 2018).
   2. HR status is defined as positive in ER expression by IHC, according to the relevant ASCO/CAP Guidelines (Allison et al. 2020)
4. Patient must have received either at least 1 year of adjuvant abemaciclib or ribociclib.
5. Recurrence of advanced breast cancer was diagnosed ≥1 year from the last dose of adjuvant CDK4/6 inhibitor.
6. Patients must have received a minimum of 2 years of adjuvant endocrine therapy (either alone or in combination with CDK4/6 inhibitors)
7. Patient has an ECOG PS 0 or 1.
8. Must have at least one measurable lesion according to RECIST v1.1. Patients without measurable lesions must have at least one lytic bone lesion.
9. Patient has adequate bone marrow and organ function as defined by the following laboratory values:

   1. Absolute neutrophil count ≥ 1.5 × 109/L
   2. Platelets ≥ 100 × 109/L
   3. Hemoglobin ≥ 9.0 g/dL
   4. Serum creatinine < 1.5 mg/dL or CCr ≥ 50 mL/day
   5. In absence of liver metastases, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) should be below 2.5 × upper limit of normal(ULN). If the patient has liver metastases, ALT and AST should be < 5 × ULN
   6. Total serum bilirubin < ULN; or total bilirubin ≤ 3.0 × ULN with direct bilirubin <1.5 x ULN of the local laboratory in patients with well documented Gilbert's Syndrome
10. Patient must be able to swallow study therapy
11. Patient must be able to communicate with the investigator and comply with the requirements of the study procedures
12. Patient must be willing to remain at the clinical site as required by the protocol.

Exclusion Criteria:

1. Patients whose cancer recurs one year or later after completing adjuvant endocrine therapy
2. Patients who have been free from endocrine therapy for at least 2 years
3. Patient whose disease recurred during or within 1 year from adjuvant CDK4/6 inhibitor treatment.
4. Patient who did receive adjuvant palbociclib irrespective of disease-free interval.
5. Patients who did not receive adjuvant CDK4/6 inhibitor treatment or who received less than 1 year of adjuvant CDK4/6 inhibitor treatment.
6. Patients who have received fulvestrant in adjuvant setting before randomization.
7. Patients who have received any line of systemic treatment for advanced breast cancer is not eligible.
8. Participant has not recovered from clinical, and laboratory acute toxicities related to prior anticancer therapies to NCI CTCAE version 4.03 Grade ≤1. Exception to this criterion: participants with grade 2 taxane-induced neuropathy, any grade of alopecia, amenorrhea or other toxicities not considered a safety risk for the participant as per investigator's discretion, are allowed to enter the study.
9. Patient has a concurrent malignancy or malignancy within 3 years of randomization, with the exception of adequately treated basal cell carcinoma, squamous cell skin carcinoma, non-melanomatous skin cancer or curatively resected cervical cancer.
10. Patient with symptomatic, unstable CNS metastases. Note: Symptomatic CNS metastases should be locally treated prior enrollment.
11. Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
12. Patient has a known history of HIV infection (testing not mandatory).
13. Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, contraindicate patient participation in the clinical study (e.g., chronic pancreatitis, chronic active hepatitis, etc.).
14. Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality, including but not limited to any of the following:

    1. History of documented myocardial infarction (MI), angina pectoris, symptomatic pericarditis, or coronary artery bypass graft (CABG) within 6 months prior to study entry
    2. Documented cardiomyopathy
    3. Long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome, or any of the following: ① Risk factors for Torsades de Pointe (TdP) including uncorrected hypocalcemia, hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia ② Concomitant medication(s) with a known risk to prolong the QT interval and/or known to cause Torsades de Pointe that cannot be discontinued or replaced by safe alternative medication (e.g., within 5 half-lives or 7 days prior to starting study drug) ③ Inability to determine the QTcF interval
    4. Clinically significant cardiac arrhythmias (e.g., ventricular tachycardia), complete left bundle branch block, high-grade AV block (e.g., bifascicular block, Mobitz type II and third-degree AV block)
15. Patient is currently receiving any of the following substances and cannot be discontinued 7 days prior to Cycle 1 Day 1:

    1. Concomitant medications, herbal supplements, and/or fruits (e.g., grapefruit, pummelos, star fruit, Seville oranges) and their juices that are strong inducers or inhibitors of CYP3A4/5
    2. Medications that have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5.
16. Patient has had major surgery within 14 days prior to starting study drug or has not recovered from major side effects of surgery.
17. Patient who has received any investigational drug(s) within 14 days prior to first day treatment or within 5 half-lives of the investigational product (whichever is longer).
18. Patient is currently receiving or has received systemic corticosteroids ≤ 2 weeks prior to starting study drug, or who have not fully recovered from side effects of such treatment.

    Note: The following uses of corticosteroids are permitted: single doses, topical applications (e.g., for rash), inhaled sprays (e.g., for obstructive airways diseases), eye drops or local injections (e.g., intra-articular).
19. Patient is concurrently using other antineoplastic agents (except for adjuvant endocrine treatment monotherapy)
20. Patient who has received radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to randomization, and who has not recovered to grade 1 or better from related side effects of such therapy (with the exception of alopecia) and/or if ≥ 25% of the bone marrow was irradiated.
21. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
22. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing of study treatment and after stopping study medication.* Highly effective contraception methods include:

    * Ribociclib : For at least 3 weeks after the last dose, Fulvestrant : For 2 years after the last dose, Everolimus : For up to 8 weeks after the last dose.

    - Effective contraception must be used as follows.
    1. Total abstinence (when this is in line with the preferred and usual lifestyle of the subject). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
    2. Total hysterectomy (surgical removal of the uterus and cervix) or tubal ligation (getting your "tubes tied") at least six weeks before taking study treatment.
    3. Male sterilization (at least 6 months prior to screening). For female subjects on the study, the vasectomized male partner should be the sole partner for that subject.
    4. Combination of the following: Barrier methods of contraception: Condom and intrauterine devices (IUDs) (e.g., loop insertion)
23. Not able to understand and to comply with study instructions and requirements.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2031-06-30 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | Up to 5 years
  From the time from randomization to first documented progression or death, whichever occurs first

SECONDARY OUTCOMES:
Overall survival | Up to 5 years
  From date of randomization to date of death due to any cause.
Objective Response Rate | Up to 5 years
  Assessed by RECIST 1.1. Cinical benefit rate defined as percentage of patients with CR, PR per RECIST 1.1 or SD lasting 24 weeks or longer
Adverse Events | Up to 5 years
  Incidence/severity of adverse events, lab abnormalities based on CTCAE4.03

IPD SHARING:
Plan to Share IPD: No